CLINICAL TRIAL: NCT03241147
Title: Interventional, Open Label, Reduced/Staged, Single Dose Study Investigating the Pharmacokinetic Properties of Lu AF35700 in Subjects With Renal Impairment and in Healthy Subjects
Brief Title: Pharmacokinetics of Lu AF35700 in Subjects With Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New data; the study was terminated based on new efficacy data
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17278A
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Lu AF35700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects with severe renal impairment (Group A) (Experimental)
  Interventions: Drug: Lu AF35700
- Healthy subjects (Group B) (Experimental)
  Interventions: Drug: Lu AF35700
- Subjects with moderate renal impairment (Group C) (Experimental)
  Interventions: Drug: Lu AF35700
- Subjects with mild renal impairment (Group D) (Experimental)
  Interventions: Drug: Lu AF35700

INTERVENTIONS:
Drug: Lu AF35700 — Single dose, 10 mg film coated tablet

SUMMARY:
This study will evaluate the pharmacokinetics of Lu AF35700 after a single dose tablet to subjects with renal impairment (kidney insufficiency) and compare that with healthy subjects

DETAILED DESCRIPTION:
If the initial data shows a substantial effect in subjects with severe renal impairment, the study will be expanded to include subjects with intermediate level (mild and moderate) of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

-Healthy subjects: The subject has a Glomerular Filtration Rate as based on creatinine clearance (CLCr) ≥90 mL/min (estimated by the Cockcroft-Gault method)

-Subjects with renal impairment: The subject has any form of renal dysfunction which includes polycystic kidney disease

The subject is classified as having renal impairment at Screening according to Cockroft-Gault method for estimating creatinine clearance:

Severe: CLCr ≤ 29 mL/min Moderate: 30 mL/min ≤ CLCr ≤ 59 mL/min Mild: 60 mL/min ≤ CLCr ≤ 89 mL/min

Exclusion Criteria:

-The subject has previously been dosed with Lu AF35700

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Predose to day 57 postdose
  Area under the Lu AF35700 plasma concentration-time curve from zero to infinity
Cmax | Predose to day 57 postdose
  Maximum observed plasma concentration of Lu AF35700

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- APEX, Munich, Germany